# Getting to Yes: Increasing COVID-19 vaccination in Michigan

Community-Centered Interventions for Improved Vaccine Uptake for COVID-19 (CIVIC)

Funded by: NIH Health and Human Services GRANT13282146 Award # 5R01MD016867-02

# National Clinical Trial (NCT) Identified #: NCT05096260

Principal Investigators: Erica Marsh. M.D. and Ken Resnicow, Ph.D.

# Approved by IRB HUM00204174

Protocol Version #: v.12.0 – February 26, 2024

| 1. | STAT | EMENT OF COMPLIANCE | |
|----|------|-------------------------------------------------------|----|
| 1 | PROT | TOCOL SUMMARY | |
| | 1.1 | Synopsis | |
| | 1.2 | Schema | 1 |
| | 1.3 | Schedule of Activities (SoA) | 6 |
| 2 | INTR | ODUCTION | 7 |
| | 2.1 | Study Rationale | |
| | 2.2 | Background | 8 |
| | 2.3 | Risk/Benefit Assessment | 8 |
| 3 | OBJE | CTIVES AND ENDPOINTS | g |
| 4 | STUE | DY DESIGN | 10 |
| | 4.1 | Overall Design | 10 |
| | 4.2 | Scientific Rationale for Study Design | 13 |
| | 4.3 | Justification for Dose | 13 |
| | 4.4 | End of Study Definition | 13 |
| 5 | STUE | DY POPULATION | 13 |
| | 5.1 | Inclusion Criteria | 13 |
| | 5.2 | Exclusion Criteria | 13 |
| | 5.3 | Lifestyle Considerations | 13 |
| | 5.4 | Screen Failures | 14 |
| | 5.5 | | |
| 6 | STUE | OY INTERVENTION | 16 |
| | 6.1 | Study Intervention(s) Administration | 16 |
| | 6.2 | Preparation/Handling/Storage/Accountability | 16 |
| | 6.2. | 1 Acquisition and accountability | 16 |
| | 6.2. | 2 Formulation, Appearance, Packaging, and Labeling | 17 |
| | 6.2. | 3 Product Storage and Stability | 18 |
| | 6.2. | 4 Preparation | 18 |
| | 6.3 | Measures to Minimize Bias: Randomization and Blinding | 18 |
| | 6.4 | Study Intervention Compliance | 18 |
| | 6.5 | Concomitant Therapy | 18 |
| | 6.5 | 1 Rescue Medicine | 18 |

| 7 STU | DY INTER | <b>VENTION DISCON</b> | TINUATION AND PARTICIPANT | |
|---|---|---|---|---|
| DISCONTIN | NUATION, | /WITHDRAWAL | | 18 |
| 7.1 | Discont | inuation of Study | Intervention | 18 |
| 7.2 | | | on/Withdrawal from the Study | |
| 7.3 | | | | |
| 8 STU | | • | OCEDURES | |
| 8.1 | | | | |
| 8.2 | | | nents | |
| <i>8.3</i> | | | us Adverse Events | |
| 8.3 | | | dverse Events (AE) | |
| 8.3 | 3.2 | | rious Adverse Events (SAE) | |
| 8.3 | 3. <i>3</i> | | f an Adverse Event | |
| | | 1.1.1.1 | Severity of Event | |
| | | 1.1.1.2 | Relationship to Study INTERVENTION | 22 |
| | | 1.1.1.3 | Expectedness | |
| 1.1 | 1.2 | Time Period an | d Frequency for Event Assessment and Follow-Up | 24 |
| 1.1 | 1.3 | | Reporting | |
| 1.1 | 1.4 | Serious Adverse | Event Reporting | 25 |
| 1.1 | 1.5 | | ts to Participants | |
| 1.1 | 1.6 | | egnancy | |
| 1.2 | Unantic | | | |
| 1.2 | | | nanticipated Problems (UP) | |
| 1.2 | 2.2 | | Problem Reporting | |
| 1.2 | 2.3 | Reporting Una | nticipated Problems to Participants | 26 |
| 2 STA | TISTICAL ( | | | |
| 2.1 | Study H | ypotheses | | 27 |
| 2.2 | Sample | Size Determinatio | on | 27 |
| 2.3 | Populat | ions for Analyses | | 27 |
| 2.4 | Statistic | cal Analyses | | 27 |
| 2.4 | 1.1 | General Appro | ach | 27 |
| 2.4 | 1.2 | Analysis of the | Primary Efficacy Endpoint(s) | 27 |
| 2.4 | 1.3 | Analysis of the | Secondary Endpoint(s) | 29 |
| 2.4 | 1.4 | Safety and Inte | rim Analyses | 29 |
| 2.4 | 1.5 | Baseline Descri | ptive Statistics | 29 |
| 2.4 | 1.6 | Tabulation of I | ndividual Participant Data | 29 |
| 2.4 | 1.7 | Exploratory An | alyses | 29 |
| 3 SUP | PORTING | <b>DOCUMENTATIO</b> | N AND OPERATIONAL CONSIDERATIONS | 29 |
| 3.1 | Regulat | ory, Ethical, and S | Study Oversight Considerations | 29 |
| 3.1 | ! <b>.1</b> | Informed Conse | ent Process | 29 |
| | | 3.1.1.1 | Consent/assent and Other Informational Documents | |
| | | | Provided to participants | 30 |
| | | 3.1.1.2 | Consent Procedures and Documentation | 30 |
| 3.1 | 1.2 | Study Discontir | nuation and Closure | 30 |
| 3.1 | 1.3 | Confidentiality | and Privacy | 30 |

| 3.1.4 | Future Use of S | tored Specimens and Data | 31 |
|---|---|---|---|
| 3.1.5 | | Study Governance | |
| 3.1.6 | Safety Oversigh | nt | 32 |
| 3.1.7 | | ring | |
| 3.1.8 | | nce and Quality Control | |
| 3.1.9 | | and Record Keeping | |
| | | Data Collection and Management Responsibilities | |
| | 3.1.9.2 | Study Records Retention | 33 |
| 3.1.10 | Protocol Deviat | ions | 34 |
| 3.1.11 | Publication and | l Data Sharing Policy | 34 |
| 3.1.12 | Conflict of Inter | rest Policy | 34 |
| 3.2 Addit | ional Considerations | | 34 |
| 3.3 Abbre | eviations | | 35 |
| 3.4 Proto | col Amend | | |
| ment Histor | y | | 35 |
| 3.5 Apper | ndices | | 2 |
| 4 REFERENCE | <u>S</u> | | 3 |
| 5 PROTOCO | L SIGNATURE PAGE | 11 | |

#### STATEMENT OF COMPLIANCE

This study will be carried out in accordance with Good Clinical Practice (GCP) as required by the following:

- United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, and 21 CFR Part 56)
- NIH Clinical Terms of Award

All key personnel (all individuals responsible for the design and conduct of this study) have completed Human Subjects Protection Training. The protocol and informed consent form(s) will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form will be obtained before any participant is enrolled. Any amendment to the protocol will first go through IRB review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be IRB-approved; a determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form, if this becomes applicable. (i.e. if there is a requested change to the consent form during the course of this study)

#### 1 PROTOCOL SUMMARY

#### 1.1 Synopsis

Title:

Getting to Yes! Michigan: Increasing COVID-19 vaccinations

Study Description:

This proposal, entitled Community-Centered Interventions for Improved Vaccine Uptake for COVID (CIVIC), is designed to directly address and decrease COVID-19 vaccine hesitancy and increase vaccine uptake among populations that experience COVID-19 related disparities. We will focus on the entirety of the state of Michigan, with a keen focus in four counties within Michigan where a disproportionate burden of COVID-19 within AA and LX communities, i.e., Wayne, Genesee, Kent and Washtenaw Counties. Using a community-based participatory research (CBPR) approach, CIVIC will leverage: its long term, community-based relationships through an established CBPR Steering Committee developed as a Community Engagement Alliance (CEAL) grant recipient, the University of Michigan CTSA (MICHR), and the expertise of our academic partners to identify and understand factors that contribute to COVID-19 vaccine hesitancy in AA and LX communities in Michigan.

**Objectives:** 

1: Increase understanding of the barriers and drivers of vaccine uptake and hesitancy;

2: Increase vaccine uptake and decrease vaccine hesitancy through the implementation and evaluation of a multilevel, tailored intervention; and maintain, enhance, and evaluate the effectiveness of the CIVIC partnerships to

equitably engage all partners.

**Endpoints:** 

<u>Primary Endpoint</u>: Vaccination rate between baseline and 6-months <u>Secondary Endpoints</u>: Vaccination rate between baseline and 12 months **Study Population:** Adults (>18-years-old) living in the state of Michigan. We have recruited 30

churches into the intervention, and they will assist in the recruitment of subjects from each church alongside study team recruitment in the community. To achieve the goal of the study, we must recruit  $n=800-1000\ (400-500)$  intervention, (400-500) control) subjects. We expect an approximately equal distribution of gender. Demographics are expected to reflect local community

populations from which we recruit.

Phase: N/A

Description of Sites/Facilities Enrolling Participants:

Will recruit subjects from the community at events such as farmers markets, health fairs, social media, etc as well as from the thirty churches from the four target counties. We will also recruit with Data Direct, a U-M resource.

Description of Study Intervention:

Intervention designed as a randomized control trial implemented over 48 weeks. Intervention includes SMS/MMS messages tailored from a Baseline survey for people who are either unvaccinated/unboosted. Volunteers who are vaccinated may participate as vaccine champions to encourage participants to be vaccinated. If the fully vaccinated person has signed up prior to December 2022, they can complete 2 trainings to become a vaccine champion plus. They will reach out to participants that would like additional information from a vaccine champion plus. A fully vaccinated person enrolled after January 2023 will become a vaccine champion and will have the opportunity to complete the motivational interviewing training but won't interact with participants.

**Study Duration:** 48 weeks for intervention and manuscript preparation time

Participant Duration:

24 weeks

Related

N/A

separate QI initiatives for this

study

#### 1.2 Schema

Crossover Individualized Randomized Control Trial

Randomization. At the time of randomization, eligible participants will be assigned a unique randomization number; no participant may begin intervention prior to randomization. Eligible participants will be randomized to Intervention or Control in a 1:1 manner, stratified by vaccination status (vaccinated [ $\geq$ 1 vaccine received] or unboosted or unvaccinated [0 vaccines received]). The study statistician will prepare the randomization schedule, using computer-generated permuted

block randomization with the block size(s) known only by the study statistician. A secure web-based application will be built that will be used by the coordinators to enter participant information (e.g., participant ID, stratification factor) and to obtain the randomization number.

#### Mock Randomization:

| Randomization List 1: | Vaccinated ( | (>1 vaccine received) |
|-----------------------|--------------|-----------------------|

| STRAT_NO | STRAT_LABEL | TRT_GROUP | TRT_ALLOCATION | RANDO_NO |
|---|---|---|---|---|
| | <del>-</del> | _ | <del>-</del> | _ |
| 1 | Vaccinated (≥1 vaccine received) | Α | Control | 1327 |
| 1 | Vaccinated (≥1 vaccine received) | Α | Control | 1330 |
| 1 | Vaccinated ( <u>&gt;</u> 1 vaccine received) | В | Intervention | 1333 |
| 1 | Vaccinated (≥1 vaccine received) | В | Intervention | 1336 |
| 1 | Vaccinated (≥1 vaccine received) | Α | Control | 1339 |
| 1 | Vaccinated ( <u>&gt;</u> 1 vaccine received) | В | Intervention | 1342 |
| 1 | Vaccinated ( <u>&gt;</u> 1 vaccine received) | В | Intervention | 1345 |
| 1 | Vaccinated ( <u>&gt;</u> 1 vaccine received) | Α | Control | 1348 |
| Randomization List 1: Unboosted or Unvaccinated (0 vaccines received) | | | | |
| Randomizat | ion List 1: Unboosted or Unvaccinated (0 <sup>,</sup> | vaccines receive | d) | |
| Randomizat<br>STRAT_NO | ion List 1: Unboosted or Unvaccinated (0) STRAT_LABEL | vaccines receive<br>TRT_GROUP | d)<br>TRT_ALLOCATION | RANDO_NO |
| | • | | • | RANDO_NO<br>1351 |
| STRAT_NO | STRAT_LABEL | TRT_GROUP | TRT_ALLOCATION | <del>-</del> |
| STRAT_NO<br>0 | STRAT_LABEL Unboosted or Unvaccinated (0 vaccines received) | TRT_GROUP<br>B | TRT_ALLOCATION Intervention | 1351 |
| STRAT_NO<br>0<br>0 | STRAT_LABEL Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) | TRT_GROUP<br>B<br>A | TRT_ALLOCATION Intervention Control | 1351<br>1354 |
| STRAT_NO 0 0 0 | STRAT_LABEL Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) | TRT_GROUP<br>B<br>A<br>B | TRT_ALLOCATION Intervention Control Intervention | 1351<br>1354<br>1357 |
| STRAT_NO<br>0<br>0<br>0<br>0 | STRAT_LABEL Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) | TRT_GROUP B A B | TRT_ALLOCATION Intervention Control Intervention Control | 1351<br>1354<br>1357<br>1360 |
| STRAT_NO<br>0<br>0<br>0<br>0<br>0 | STRAT_LABEL Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) Unboosted or Unvaccinated (0 vaccines received) | TRT_GROUP B A B A | TRT_ALLOCATION Intervention Control Intervention Control Intervention | 1351<br>1354<br>1357<br>1360<br>1363 |

Primary Outcome: Primary outcomes will be **vaccine completion** ((2mRNA or 1 J & J) + bivalent) Secondary Outcome: Primary outcome is **additional vaccine dose** (0 to 1, 1 to 2, or 2 to 3)

We aim to enroll around 500 per arm (moderate effective size e.g., 20% vs. 32% rates in control vs. intervention arms).

#### 1.3 Schedule of Activities (SoA)

Note: Times indicated in this table guide our study measures and time points. Our pilot work has shown that patient scheduling for activities requires flexibility to accommodate not only the study but the needs and schedules of patients. As such, times for data collection may show 'windows +/- x days). Exact time points of data collection will be documented in study logs, and also accounted for during analyses.

| Pre | Post |
|-----|------|
|-----|------|

| Event-Time Point | Baseline | Follow-up |
|--------------------------------------------|----------|-----------|
| Church Enrollment | Х | |
| Individual Enrollment | Х | |
| Baseline for unvaccinated | Х | |
| Virtual training for recruited champions | Х | |
| In-person training for recruited champions | Х | |
| Post-intervention Survey | | х |

#### 2 INTRODUCTION

# 2.1 Study Rationale

Like many states across the country, COVID-19 cases and deaths have impacted communities of color in Michigan at disproportionately higher rates than whites. A staggering reality is that while African Americans (AA) represent only 13.6% of Michigan's population, they represent 40% of the deaths from COVID-19.

- Half of the cases and deaths in Michigan occurred in Wayne County.
- Other Counties in the lower half of Michigan have similar disparities including Genesee, Washtenaw, and Kent.
- - In Genesee County, where AAs represent 20.3% of the population, they represent 35% of COVID-19 cases and 45% of deaths.
- -- In Washtenaw County, nearly half of the cases to date are located in two majority low-income zip codes in the city of Ypsilanti. AA residents, who make up 12% of the Washtenaw population, disproportionately constitute more than a quarter of the cases.
- -- And in Kent County, while 10.8% of the population is Latinx (LX), this ethnic group makes up 32.4% of COVID-19 cases.

Preliminary data from the state reveal that these disparities will likely worsen due to significant hesitancy, fear, mistrust and misinformation regarding the COVID-19 vaccine if nothing is done to change current trends. This proposal, entitled Community-Centered Interventions for Improved Vaccine Uptake for COVID-19 (CIVIC), is designed to directly address and decrease COVID-19 vaccine hesitancy and increase vaccine uptake among populations that experience COVID-19 related disparities.

CIVIC/G2YMI will be offered to anyone in the state of Michigan, we will focus on the four counties within Michigan where a disproportionate burden of COVID-19 is within AA and LX communities, i.e., Wayne, Genesee, Kent and Washtenaw Counties. Using a community-based participatory research (CBPR) approach, CIVIC will leverage: its long term relationships with the communities involved, an established CBPR Steering Committee developed and the knowledge gained as a Community Engagement Alliance (CEAL) grant recipient, the resources and networks of the University of Michigan CTSA (MICHR), and the

expertise of our academic partners to identify and understand factors that contribute to COVID-19 vaccine hesitancy in AA and LX communities in Michigan.

This aim will develop and test interventions based on community-centered approaches to achieve a primary goal of increased vaccine uptake.

We will achieve this goal with the following aims:

- 1: Increase understanding of the barriers and drivers of vaccine uptake and hesitancy;
- 2: Increase vaccine uptake and decrease vaccine hesitancy through the implementation and evaluation of a multilevel intervention; and maintain, enhance, and evaluate the effectiveness of the CIVIC partnership to equitably engage all partners.

#### 2.2 Background

Like many states across the country, COVID-19 cases and deaths have impacted communities of color in Michigan at disproportionate rates. A staggering reality is that while African Americans represent only 13.6% of Michigan's population, they represent 40% of the deaths from COVID-19. Half of the cases and deaths in Michigan occurred in Wayne County. Other Counties in the lower half of Michigan have similar disparities including Genesee, Washtenaw, and Kent. In Genesee County, where African Americans represent 20.3% of the population, 35% of COVID-19 cases and 45% of deaths are in these communities. In Washtenaw County, nearly half of the cases to date are located in two majority low-income zip codes in the city of Ypsilanti. African American residents, who make up 12% of the Washtenaw population, disproportionately constitute more than a quarter of the cases. And in Kent County, while 10.8% of the population is Hispanic or Latino, this ethnic group makes up 32.4% of COVID-19 cases. It is unquestionable that this crisis has exacerbated existing racial/ethnic inequity and health disparities in Michigan. Preliminary data from the state reveal that these disparities will likely worsen due to significant hesitancy, fear, mistrust, and misinformation regarding the COVID-19 vaccine if nothing is done to change current trends. This proposal, entitled Community-Centered Interventions for Improved Vaccine Uptake for COVID (CIVIC) is designed to directly address and decrease COVID-19 vaccine hesitancy and increase vaccine uptake among populations that experience health disparities. We will focus on the four counties within Michigan that were hardest hit and/or where a disproportionate burden is within AA and LX communities i.e., Wayne, Genesee, Kent and Washtenaw Counties. Using a community based participatory research (CBPR) approach, CIVIC will leverage its long term relationships with the community, an established Steering Committee, the resources and networks of the University of Michigan CTSA (MICHR), our status and knowledge gained as a Community Engagement Alliance (CEAL) grant recipient, and the expertise of our academic partners to identify and understand factors that contribute to COVID-19 vaccine hesitancy in African-American (AA) and Latinx (LX) communities in Michigan and develop and test interventions based on community-centered approaches to achieve a primary goal of increased vaccine uptake.

# 2.3 Risk/Benefit Assessment

<u>Risk Likelihood:</u> There is the rare potential risk that participants may be embarrassed or upset by questions in the questionnaires or interviews. Risks or discomforts from this research are minimal and may include discomfort with speaking to unvaccinated individuals about their barriers and beliefs about the COVID-19 vaccine.

<u>Risk Seriousness:</u> You have the option to not answer any questions that you feel is too sensitive. Questions were previewed by community members, religious and spiritual leaders, and those questions deemed too sensitive were removed.

<u>Measures to minimize risk:</u> Privacy is very important, and the study investigators use many safety measures to protect subject privacy.

Participation in this research is voluntary, and you may choose to withdraw at any time by contacting the study team at <a href="mailto:gettingtoyesMl@med.umich.edu">gettingtoyesMl@med.umich.edu</a>

Participation in this research is confidential. All research data will be de-identified, and you will be identified by number and not by name. No information by which you can be identified will be released or published in connection with this study.

No information by which you can be identified will be released or published in connection with this study. In spite of all of the safety measures that we will use, however, we cannot guarantee that your identity will never become known.

Study paper data (i.e. consent forms and history forms will be stored in locked cabinets) and electronic data is stored on servers accessible via password-protected computers.

Study data will be stored in a relational database on a separate highly restricted secure server. Databases will be backed up daily to an offsite NAS storage device using automatic backup software that is available 24/7 except for scheduled maintenance. Only the primary investigators and other authorized research team members named in the approved IRB application will have access to the de-identified data. These standards will help ensure that violations of confidentiality will be minimal.

There is the potential risk that participants may be embarrassed or upset by questions in the questionnaires or interviews. Subjects will have the option to not answer any questions that they determine to be too sensitive.

The direct benefits of your participation may include:

- increased knowledge about the COVID-19 vaccine.

There are no immediate health benefits to the study subjects. This study, however, will provide important information about the beliefs, behaviors, sources of truth, and misinformation that drive COVID-19 vaccine uptake so that in the future others might benefit from this study.

Participants who wish to receive communication training will receive a link to the Articulate 360 training. Newly Enrolled (Post December 2022) Vaccine Champions will complete the virtual, MI-based, (Articulate) communications training only. No incentive will be paid to newly enrolled Vaccine Champions. Note: Currently enrolled (prior to December 2022) Vaccine Champions Plus will be trained on program specifics to aide in discussions with participants to answer questions regarding vaccination. They will receive abbreviated PEERRS training as well as Motivational Interviewing techniques. We will distribute vaccine champions plus initial \$50 payment after a self-paced virtual and \$50 for a live-virtual MI-based communication trainings.

Vaccine Champions Plus (those recruited prior to Dec 22) will be matched manually to unvaccinated/unboosted participants manually by the study team.

Link to Articulate Training: <a href="https://rise.articulate.com/share/U3TRBPxQQKA5Vd8yOs4w6aVOtuq-FKyJ">https://rise.articulate.com/share/U3TRBPxQQKA5Vd8yOs4w6aVOtuq-FKyJ</a>

#### 3 OBJECTIVES AND ENDPOINTS

- 1: Increase understanding of the barriers and drivers of vaccine uptake and hesitancy;
- 2: Increase vaccine uptake and decrease vaccine hesitancy through the implementation and evaluation of a multilevel intervention; and
- 3: Maintain, enhance, and evaluate the effectiveness of the CIVIC partnership to equitably engage all partners.

#### 4 STUDY DESIGN

#### 4.1 Overall Design

Overview and Study Design.

We will develop and test, with the active engagement of the CIVIC SC, the impact of a tailored mobile-optimized web intervention on vaccine uptake. Individually tailored interventions have consistently been shown to be more efficacious than group-level or static messages.

Building on several prior individually-tailored interventions we have developed for AAs, we designed a user-friendly, culturally-sensitive, interactive intervention that addresses key determinants of vaccine behavior—e.g., knowledge gaps, barriers, beliefs, values, ethnic identity, medical mistrust, discrimination, and communal responsibility. The comparison group will receive a mobile-optimized web program absent individual tailoring (i.e., standard, static content). Participants, (unboosted or unvaccinated) will be randomly assigned to each condition, for both Aims 2 and 3. The primary outcome will be self-reported COVID-19 vaccine uptake (at least one dose) after six months from the start of the Aim 2 study. To detect a 15% absolute difference in vaccine rates (.40 versus .55), we will require approximately 700 individuals at posttest (350 from intervention, 350 from control)

All intervention materials are available in English and Spanish including: the web-based program messages through testimonials, infographics, and links to other content, promotional materials.

#### App Structure.

The "App," which will be web-based rather than a native program running in iOS or Android, will be optimized for use with various screen sizes, devices, and operating systems. This allows us to avoid the time and cost of developing and posting native versions in iOS/Swift and Android. To allow use across multiple device types (e.g., phone, PC, or tablet) without requiring participants to download an actual "App." The mobile website is a hybrid, meaning that it is neither a truly native mobile application (because much of the computation is done via the web) nor purely web-based. Our team has built numerous similar sites and has extensive experience with Qualtrics, Cordova, CSS, HTML, Python, and Java, including projects by Drs. Resnicow and An. Users will "download" and bookmark the "App" which will "launch" upon clicking, mimicking a true App experience.

#### App Development.

The Center for Health Communications Research (CHCR), which will design the tailored web program for this study, has been at the forefront of theory-driven, culturally-tailored interventions for over 20 years. CHCR iteratively evaluates and improves the user experience throughout the development process, relying on a range of feedback methods including contextual interviews, focus groups, heuristic evaluation, and formal usability testing conducted in accordance with best practices outlined at usability.gov. As part of the project lifecycle, CHCR performs qualitative and quantitative evaluation of user experience with mature programs (e.g. system usability and paradata assessment) and the impact of user experience on intervention impact. A robust and refined project lifecycle, based on quality principles and modern agile development methodologies, guides all planning, development, and implementation activities. This standard process helps ensure well-conceived, high-quality products by defining goals, methods, and quality assurance procedures for each of the project's stages. CHCR uses a standards-based, cross-platform, open-source application that enables the efficient creation, testing, and delivery of richly tailored communications. These communications may include individually-tailored

text and media (photos, graphics, animations, audio, video) delivered via a range of channels. Because of the common technical platform, resulting in tailored programs are easier to disseminate.

#### Theoretical Framework.

Our primary framework that will guide the web content is Self-Determination Theory (SDT). SDT differentiates between autonomous and controlled behavioral regulation. Behaviors are autonomous when they result from conscious choice and are personally relevant. Conversely, behaviors are considered controlled when performed due to pressure or coercion, either by external or internal forces. A key principle of SDT is that messages that enhance autonomy and perceived competence and are consistent with a person's values and goals will be more effective in changing behavior than messages focusing on external rewards such as pleasing others, fear of disease, or avoiding guilt, anxiety, or shame. To link vaccination to broader values and goals, in the baseline assessment, participants will be presented with approximately 20 values/life goals, from which they will select 3-4 goals that are important to them; individually tailored messages will link each of these values to vaccination. For example, if an individual chooses family or strength as key values, we will provide messages that link vaccination to being there for their family or to remain independent. We will also tailor testimonials based on member values and communication style preference (see below). Another component of autonomy that is relevant here is providing choice as to how much and what information participants receive.

## Individual-Level Tailoring Message Content.

CHCR will tailor the content based on key determinants of vaccine behavior including knowledge, barriers, benefits/drivers, cultural values, mistrust, ethnic identity, communication preferences, and the personal meaning of vaccination. The final list for tailoring content will be determined by our Aim 1 formative research, preliminary data collected as part of our C3 study, and analysis of other sources. The CIVIC SC will play a critical role in reviewing these materials and deciding on the final list of content for tailoring. The mobile-optimized website will include a brief assessment of these constructs, generally using measures we have already developed. Using other methods such as testimonials, we will deliver individualized content addressing each of these constructs. For example, for someone who reports they are worried about contracting the virus from the vaccine, we will offer them what we call "essential facts" about the topic and then provide "drill down" options if they want to learn more. We will also tailor messages to drivers that we know are primary for the COVID-19 vaccine: communal responsibility and individual choice/personal health protection. For example, for someone high on communal responsibility, we will reflect this back to them in their message as "... if you got vaccinated, you would feel you are protecting others in your community..." or "... how will you feel about being a leader in your community by getting vaccinated?" Similarly, someone high on individual choice/personal health protection will be provided with feedback such as "getting the vaccine is a personal choice for you, not something you want to be shamed or pressured into doing." Similar tailored messages will be developed for each of the target mediators.



# How we will deliver messages:

- Collect baseline answers to assess concerns
- Feed baseline data into system code to determine:
  - a) Appropriate tailored message (where able)
  - b) Optimal message delivery order
- 3) Text messaging system delivers tailored content first, targeted info second

AAs are heterogeneous with regard to racial identity and this variability should be considered when designing health messages and programs for AAs. We have demonstrated that for AAs whose racial identity is central to their overall identity, messages that refer to or link race to the target behavior can be highly salient. However, for AAs with low racial centrality, framing messages around race can be poorly received or even harmful. Thus, we will use our brief message of racial centrality, based on the work of Sellers, to classify individuals by their ethnic identity and deliver messages differentially framed on respondents' identity. For example, for those with high racial centrality, we would frame their message as "... getting the vaccine can help protect other AAs from getting COVID" or "AAs have a higher rate of COVID than other Americans." For those with low racial salience, we would frame the message as "... getting the vaccine can help protect other Americans from getting COVID" or "Americans have a higher rate of COVID than other countries."

Individual-Level Tailoring Message Tone.

In several prior studies, we found that message tone impacts uptake. We have developed a tailoring algorithm that optimizes message tone based on communication preference. We assess preference with two items, one assessing the global trait preference and the other assessing preferences related to vaccine uptake. The trait item will be: "In general, when it comes to my health I would rather an expert just tell me what I should do." The state item will be: "When it comes to getting a COVID-19 vaccine I would rather an expert just tell me what I should do".

The two preference styles, which we call PUSH (directive) and PULL (autonomy-supportive), receive different tone, language, and content. The PULL tone uses more tentative and autonomy-supported language, whereas the PUSH tone is more definite and directive. Specifically, individuals preferring the PUSH style will be provided with directive advice describing what they "should do" regarding COVID-19 vaccination. Individuals preferring the more autonomy-supportive PULL tone will receive more tentative language such as "might" or "can," using questions (e.g., "How might you feel about getting the vaccine?" versus "You will feel good about yourself if you get the vaccine") and suggestions more than commands, helping them find personal meaning to make a vaccination decision.

App Usage

Champions are vaccinated persons from participating counties, who agree to consent to the study, and receive Motivational Interviewing Training to communicate with community members about their motivators and barriers to receiving the COVID-19 vaccine. Champions may join the study as vaccinated persons, or if previously enrolled as an unvaccinated participant, can become a Champion once vaccinated.

## 4.2 Scientific Rationale for Study Design

Aims 2 and 3 uses an individually randomized design spanning 6-months. This greatly improves the feasibility of the study as our community partners strongly encouraged us to allow all participants to receive the social marketing and Champions interventions without much delay.

Secondary outcomes include Vaccine Intentions, a continuous variable.

Participants who were unvaccinated or unboosted at will receive the intervention after completing follow-up at six months. This cohort will be followed until they are vaccinated or until the end of the study, six-months after follow-up of the primary intervention.

# 4.3 Justification for Dose

1 vaccine from baseline survey

# 4.4 End of Study Definition

At the end of the intervention period following the completion of follow-up survey. PHI will be stripped, data will be deidentified.

#### **5 STUDY POPULATION**

#### 5.1 Inclusion Criteria

Eligibility inclusion criteria:

- unvaccinated and unboosted adults 18 years and older who are interested in participating in the study
- Must be able to read and write in English or Spanish
- Must be able to receive SMS/MMS/text messages

#### 5.2 Exclusion Criteria

Exclusion criteria:

- Persons under the age of 18
- unable to read or write English or Spanish
- unable or unwilling to receive SMS/MMS
- unwilling to consent
- for vaccine champions-unwillingness to complete communication trainings in English

No specific racial, ethnic, nor gender group is excluded.

#### 5.3 Lifestyle Considerations

Not applicable.

#### 5.4 Screen Failures

- Persons under the age of 18
- unable to read or write English or Spanish
- unable or unwilling to receive SMS/MMS
- unwilling to consent
- -for vaccine champions-unwillingness/unable to complete communication trainings in English

# 5.5 Strategies for Recruitment and Retention of Participants

- 1) Change in recruitment procedures or documentation.
  - a. Recruitment will be expanded to allow all Michiganders to enroll.
  - b. In addition to recruiting from churches, we will expand enrollment to public events and forums such as attending health fairs, community baby showers, farmers markets, bus stops, social media, online blogs, etc.
  - c. After Ame00138260, Recruitment expanded to include Data Direct
    - i. Individuals meeting eligibility criteria from DataDirect will be contacted by phone, up to 8 times over a 6-week period. Recruiters will use the script in "8.1-6\_AME00138260\_HUM00204174\_Data-Direct-Recruitment-Script\_English.pdf(0.01)" or
    - 6\_AME00138260\_HUM00204174\_Data-Direct-Recruitment-Script\_English.pdf(0.01)" or "8.1-6\_AME00138260\_HUM00204174\_Data-Direct-Recruitment-
    - Script\_Spanish.pdf(0.01)" as appropriate. Individuals will be contacted by IRB-approved study team members from the study's phone # (734) 615-2860. Individuals identified as meeting eligibility criteria from DataDirect will be included in a file sent securely to the G2YMI study team. File data elements include name, phone, email. While vaccination status is not included in the file, only individuals who are not currently up-to-date, according to their MiChart EMR, will be provided to the study team, and contacted to invite to participate.
- 2) If someone is interested in participating they may enroll at www.g2ymi.org ("the website"). The electronic survey and responses are stored on secure servers. They may access this URL by:
  - a. type "the website" into an internet browser or
  - b. request a link to "the website" be sent to them via SMS (data and service charges may apply depending on a person's phone carrier and plan)
  - c. receive the link in their secured inbox in their U-M Health Research account
  - d. Receive the link by phone.

Newly Enrolled (post December 2022) Vaccine Champions will complete the virtual, MI-based, (Articulate) communications training only. No incentive will be paid to newly enrolled Vaccine Champions. Note: Currently enrolled (prior to December 2022) Vaccine Champion Plus will be trained on motivational interviewing and COVID-19 vaccine facts. They will receive abbreviated PEERRS training as well as Motivational Interviewing techniques. We will distribute vaccine champions initial \$50 payment after a self-paced virtual and \$50 for a live-virtual MI-based communication training.





Privacy is critical to the study team and steps to maintain confidentiality of research subjects is described in Section 6 of this application.

Neither participant information, nor consent/enrollment status, will not be shared with any participants' healthcare providers.

P.I. Dr. Ken Resnicow and Co-I Pastor Williams meets with RSL from the four intervention counties, who meet on a monthly basis, and will decrease as the study continues. All RSL from the counties are invited and encouraged to attend the meetings, along with study team members. These meetings are currently virtual.

#### **6 STUDY INTERVENTION**

#### 6.1 Study Intervention(s) Administration

MI Training for Champions the digital version can be found here.

https://360.articulate.com/review/content/1b8f6140-026e-4ee8-91b7-419bdc3cf7c3/review SMS/MMS Intervention

**Human Subjects Training for Vaccine Champions** the digital version can be found here. https://docs.google.com/presentation/d/1t2SD4gAPkggBPTwRbByaXxPVKoPDt2NsbAWnPEiT8gA/edit?usp=sharing

# 6.2 Preparation/Handling/Storage/Accountability

#### 6.2.1 Acquisition and accountability



6.2.2 Formulation, Appearance, Packaging, and Labeling

# The Participant Experience: Website

The participant will go to www.g2ymi.org to enroll in the program

Their view of the website will vary based on data captured during enrollment:

- Vaccination Status
- · Control vs. Intervention Status
- Content created for churches/communities (if applicable)









# 6.2.3 Product Storage and Stability

Not applicable

#### 6.2.4 Preparation

Not applicable

## 6.3 Measures to Minimize Bias: Randomization and Blinding

Using an individual-randomized design and working through the same churches (AA only) that participated in the Aim 2 multilevel intervention, we will develop and test, with the active engagement of the CIVIC SC, the impact of a tailored mobile-optimized web intervention on vaccine uptake. Individually tailored interventions have consistently been shown to be more efficacious than group-level or static messages. Participants, none of whom will have been vaccinated, will be randomly assigned to each condition.

# 6.4 Study Intervention Compliance

We are not anticipating any AE's. We are collecting limited data from subjects. Routine study monitoring by the PMs and technology staff at CHCR, could identify a reportable event, such as concerns following the approved protocol, IRB application, or agreements with the NIH and this award. Unexpected adverse events (i.e., has NOT been addressed or described in one or more of the following: Informed consent document(s) for this study, IRB application for this study, grant application or study agreement, protocol or procedures for this study, investigators' brochure or equivalent (for FDA regulated drugs or devices), DSC Reports, published literature, other documentation)

# 6.5 Concomitant Therapy

Not applicable.

#### 6.5.1 Rescue Medicine

Not applicable.

# 7 STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 7.1 Discontinuation of Study Intervention

Previously collected data will remain intact, until the end of the intervention collection period when it's deidentified. No further contact or data collection will occur.

#### 7.2 Participant Discontinuation/Withdrawal from the Study

While the study team does not anticipate the need to end a subject's participation, nor a Champion's participation, they will routinely monitor and review the study for adverse events (AE) or other reportable events such as protocol deviations (ORIO). Unexpected, clinically significant, findings will be reported as an AE/ORIO with this application.

Should a participate request withdraw, the study team member will follow-up with the participant, unless requested not to be contacted, to assess a possible reportable event.

If a Champion is found to disseminate information in contradiction to the information provided with their MI training or the CDC recommendations, they may be corrected and offered an opportunity for improvement or be asked to stop their participation.

#### 7.3 Lost to Follow-Up

Participants who have not been reached for at least 8-weeks after enrollment, or about 10 times for recruitment, will be considered lost to follow-up. Participants may resume the intervention at the point they left off.,

#### 8 STUDY ASSESSMENTS AND PROCEDURES

#### 8.1 Efficacy Assessments

#### **Eligibility:**

- unvaccinated/unboosted adults 18 years and older who are interested in participating in the study
- Must be able to read English or Spanish
- Must be able to receive SMS/MMS/text messages

**Screening:** Community members who text to enroll will receive an SMS/MMS with a link to complete eligibility screening and consent.

- Unvaccinated/unboosted enrollees may enroll in the SMS/MMS intervention.
- Fully Vaccinated individuals may become Vaccine Champions for their community. Prior to December 2022, those that are enrolled will become Vaccine Champion Plus and were primarily recruited through the collaborating churches. VC+ will complete the Motivational Interviewing (MI) Training, which provides evidence-based methods to communicate about motivators and barriers to health interventions, over Zoom, if in-person activities are not permitted at the time of the training. At the MI Training, Champions will be informed of how to assess when the person might need follow-up to discuss their barriers and motivators for the vaccine. VC+'s will be manually matched to participants by the study team. They will have access to identifiable information through the G2YMI dashboard under the vaccine champion permissions on G2YMI.

-After January 2022, fully vaccinated individuals can become vaccine champions. They will not interact with participants. The champions can complete the Motivational Interviewing training on the Articulate 360 platform.

# Recruitment and study procedures:

RSL will agree to recruit their church attendees by completing the via one church-wide announcement using the communication method preferred by their congregation (i.e face-to-face, phone, email) using the Key Facts Script that includes the URL and QR code to the Eligibility Screener and Consent.

We will also work with the CIVIC Steering Committee (SC) for recruitment of individuals in the four focal communities. The SC is made up of community leaders from across Wayne, Washtenaw, Genesee and Kent counties.

Previous to the RCT change, we enrolled church RSL who expressed interest in participating by completing the survey located in 10-1.6 Church-Eligibility-Survey\_HUM00206580. Recipients of the survey will be encouraged to distribute the survey to their own networks to reach the eligible churches. We will continue to work with the RSL and staff from our 32 collaborating churches.

- Survey data collection is done using Qualtrics (baseline, check-in, 6mo follow-up). We use the instance of Qualtrics under the UM license which is approved for collection of sensitive data.
- Electronic signatures are obtained for CIA and PPA forms using SignNow. Potential Enrollees who text to enroll will receive an SMS/MMS with a link to complete eligibility screening and consent.
  - SMS/MMS are sent via Twilio.
  - Unvaccinated/unboosted enrollees may enroll in the SMS/MMS intervention
  - Vaccinated enrollees
- Enrolled prior to Dec 2022, may become vaccine Champions for their community. Champions will complete the Motivational Interviewing (MI) Training, which provides evidence-based methods to communicate about motivators and barriers to health interventions, over Zoom, if in-person activities are not permitted at the time of the training. At the MI Training, Champions will be informed of how to assess when the person might need follow-up to discuss their barriers and motivators for the vaccine. Human subjects in research training will also be provided.
- Enrolled after Dec 2022, may complete the MI (Articulate) online training to aid conversations around vaccine hesitancy but will not interact with participants.

We will be recruiting people at community events and locations such as health fairs and bus stops. We will also utilize social media in our recruitment efforts. We will be using face-to-face communications, scripts (attached) and other recruitment materials such as flyers, posters, business cards.

Recruitment of those from Data Direct will contact individuals using IRB-approved phone scripts (attached in eResearch 08-1).

#### 8.2 Safety and Other Assessments

A Data Safety Committee (DSC) will be put into place as an integral part of the study's manual of procedures—to monitor participant safety and evaluate the ability of the investigators to conduct the proposed study with utmost regard for participant, Champion, and church protection and confidentiality. The study will not begin without approvals of the University of Michigan IRB. The PI and study team will conduct periodic reviews of regulatory requirements.

In addition, in accordance with federal regulations, the Data Safety Committee will convene to act in an advisory capacity to the study and NIH NIDDK to monitor patient safety and evaluate the ability of the investigators to conduct the proposed research with utmost regard for patient protection and confidentiality. The DSC will undertake the following tasks:

- 1. Approve initiation of the proposed study prior to study enrollment.
- 2. Review the research protocol, informed consent documents, and plans for data safety and monitoring.

3. Evaluate the progress of the study including periodic assessments of data quality and timeliness, participant recruitment, accrual and retention, participant risk versus benefit, performance of the clinical centers, and other factors that may affect study outcomes. This will occur on an ongoing basis.

- 4. Consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on the safety of the participants or the ethics of the study.
  - 5. Protect the safety of the study participants.
  - 6. Report on the safety and progress of the study.
- 7. Make recommendations to the study team and NIH HHS, and if required, to the IRBs concerning continuation, termination or other modifications of the study based on the observed beneficial or adverse effects of the study procedures.
- 8. Review interim analysis in accordance with stopping rules that will be developed for the study protocol and that will be defined in advance of data analysis and have approval of the DSC.
  - 9. Ensure the confidentiality of the study data and the results of monitoring.
- 10. Assist the funding agency by commenting on any problems of study conduct, enrollment, sample size, and/or data collection.

All aspects of the proposed research will be conducted with utmost regard for the welfare and privacy of the volunteer participants. The DSC meetings shall be closed to the public because discussions may address confidential patient data. Urgent or emergent meetings of the DSC may be called at any time or in the event of issues regarding patient safety. The format for the DSC meetings may be open or closed as dictated by the agenda of the meeting.

Termination of the Study: A majority vote of the DSC will be required to issue a study termination recommendation. Potential reasons could be but are not limited to:

- 1. An exceedingly large number of serious and unexpected adverse events.
- 2. Severe and not rectifiable logistical or data quality problems.

The DSC will consist of study team members who include a clinical leader and well-established researcher, PMs, Research Assistants, and the PI. The study biostatistician will be available to provide input and/or attend the DSC meetings, as needed.

In addition, any data integrity and patient safety-related issues will be prioritized. At study start, all research personnel, coaches and staff will undergo training and in-service meetings about study procedures. The importance of data security and compliance with procedures will be emphasized. All study personnel are required to complete and be certified by the Program for Education and Evaluation in Responsible Research and Scholarship (PEERRS) at the University of Michigan every 3 years (or equivalent, i.e. CITI training as applicable depending on University/site affiliation). A standard reporting form for adverse events will be created and completed by study personnel on an as-needed basis. Adverse events will be discussed at biweekly team meetings or sooner if needed and reported to the IRB. Documentation of completion of tasks and DSC activities will available in the team meeting minutes and ORIO/AEs submitted to the IRB.

A Regulatory and Compliance Dropbox folder will also contain all communications to the IRB, including the initial application, study protocol, any amendments, annual IRB renewal, IRB approvals, and a summary of adverse events. It will be the responsibility of the project team to maintain and update the folder. In addition, the Project Manager/Coordinator will review consent forms, and source data at regular intervals along the study, with reviews documented in a Monitoring Log, accompanied by a Monitoring Report, which will be filed in the Regulatory Binder.

Lastly, this project includes an applicable clinical trial registered with ClinicalTrials.gov, NCT#05096260.

#### 8.3 Adverse Events and Serious Adverse Events

#### 8.3.1 Definition of Adverse Events (AE)

According to the UM Medical School Office of Research definition, an adverse event (AE) is any experience or abnormal finding that has taken place during the course of a research project and was harmful to the subject participating in the research, or increased the risks of harm from the research, or had an unfavorable impact on the risk/benefit ratio.

#### 8.3.2 Definition of Serious Adverse Events (SAE)

An adverse event (AE) or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

#### 8.3.3 Classification of an Adverse Event

#### 1.1.1.1 Severity of Event

According to the UM eResearch definition, adverse events are categorized according to the following grading system:

- 0 No adverse event
- 1 Mild AE No treatment needed
- 2 Moderate AE Resolved with treatment
- 3 Severe AE Inability to carry on normal activities, required professional medical attention
- 4 Life-threatening or disabling AE
- 5 Fatal AE

#### 1.1.1.2 Relationship to Study INTERVENTION

We will use the following levels of relationship to study intervention, which is in accordance to eResearch:

Definitely Related – There is clear evidence to suggest a causal relationship, and other possible
contributing factors can be ruled out. The clinical event, occurs in a plausible time relationship
to study intervention administration and cannot be explained by concurrent disease or other

drugs or chemicals. The response to withdrawal of the study intervention (dechallenge) should be clinically plausible.

- Probably Related There is evidence to suggest a causal relationship, and the influence of other
  factors is unlikely. The clinical event occurs within a reasonable time after administration of the
  study intervention, is unlikely to be attributed to concurrent disease or other drugs or
  chemicals.
- Possibly Related There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related", as appropriate.
- Unlikely to be related A clinical event, including an abnormal laboratory test result, whose temporal relationship to study intervention administration makes a causal relationship improbable (e.g., the event did not occur within a reasonable time after administration of the study intervention) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical condition, other concomitant treatments).
- Not Related The AE is completely independent of study intervention administration, and/or
  evidence exists that the event is definitely related to another etiology.

#### 1.1.1.3 Expectedness

The principal investigator will be responsible for determining whether an adverse event (AE) is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study intervention.

- Psychosocial difficulties
  - Potential expected and unexpected risks will be outlined for patients in the informed consent document(s).
- Potential Benefits
  - There are no immediate health benefits to the study subjects. This study, however, will
    provide important information about the beliefs, behaviors, sources of truth, and
    misinformation that drive COVID-19 vaccine uptake so that in the future others might
    benefit from this study. The risks of the study are considered minimal.
- Potential Risks
  - Likelihood: There is the "rare" potential risk that participants may be embarrassed or upset by questions in the questionnaires or interviews.
  - Seriousness: We anticipant <1% risk as subjects will have the option to not answer any
    questions that they determine to be too sensitive. Questions have been previewed by
    community members, religious and spiritual leaders, and items deemed too sensitive
    were removed from the intervention, and not listed in this application.</li>
  - Measures to minimize risk: Privacy is very important, and the study investigators will use many safety measures to protect subject privacy.
  - Participation in this research is voluntary, and they may choose to withdraw at any time by contacting the study team at <a href="mailto:qettingtoyesmi@med.umich.edu">qettingtoyesmi@med.umich.edu</a>
  - Participation in this research is confidential. All research data will be de-identified, and subjects will be identified by number and not by name. No information by which the subject can be identified will be released or published in connection with this study.

- No information by which the subject can be identified will be released or published in connection with this study. In spite of all of the safety measures that we will use, however, we cannot guarantee that subject identity will never become known.
- Study paper data i.e. consent forms and history forms will be stored in locked cabinets, and electronic data will be stored servers accessible via password-protected computers.
- Study data will be stored in a relational database on a separate highly restricted secure server. Databases will be backed up daily to an offsite NAS storage device using automatic backup software that is available 24/7 except for scheduled maintenance. Only the primary investigators and other authorized research team members named in this application will have access to the de-identified data. These standards will help ensure that violations of confidentiality will be minimal.
- The procedures outlined in this proposal are considered minimal risk. There are no anticipated medical risks.
- There is the potential risk that participants may be embarrassed or upset by questions in the questionnaires or interviews. Subjects will have the option to not answer any questions that they determine to be too sensitive.

The definitions from eResearch on expectedness is as follows:

- Unexpected adverse events (i.e., has NOT been addressed or described in one or more of the
  following: Informed consent document(s) for this study, IRB application for this study, grant
  application or study agreement, protocol or procedures for this study, investigators' brochure or
  equivalent (for FDA regulated drugs or devices), DSC Reports, published literature, other
  documentation)
- Expected adverse events (i.e., has been addressed or described in one or more of the following: Informed consent document(s) for this study, IRB application for this study, grant application or study agreement, protocol or procedures for this study, investigators' brochure or equivalent (for FDA regulated drugs or devices), DSC Reports, published literature, other documentation, or characteristics of the study population)
- This study is minimal risk and we anticipate an increased uptake in the COVID-19 vaccine in the four target counties. This will help reduce the spread of COVID-19 virus and associated misinformation.

# 1.1.2 Time Period and Frequency for Event Assessment and Follow-Up

The occurrence of an adverse event (AE) or serious adverse event (SAE) may come to the attention of study personnel during interviews of a study participant presenting for medical care, or upon review by a study monitor.

All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate case report form (CRF). Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

The study team will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Events will be followed for outcome information until resolution or stabilization.

# 1.1.3 Adverse Event Reporting

We will report all adverse event according to the UM Medical School Office of Research reporting timetable:

# Standard Adverse Event Reporting Guidelines for INTERNAL AEs Occurring at UM

This chart is for studies following IRBMED standard AE reporting and requiring CR. It may be appropriate for some studies to consider a <u>Study Specific AE Reporting Plan</u>. See the gray boxes for information about External AE and UaP reporting.

| | RELATED UNRELATED | |
|---|---|---|
| UNEX | Potential Unanticipated Problems (UaPs) <sup>3</sup> Serious Adverse Event <sup>1</sup> – resulting in • Death • Life-threatening outcome Submit AE/ORIO report as <u>soon as possible</u> , but <u>within 7 calendar</u> days of becoming aware of event. Assess SAE to determine if UaP (see below for UaP criteria). | Serious Adverse Event¹- resulting in Death Life-threatening outcome Report in aggregate form via separate AE/ORIO submission in conjunction with SCR. |
| P<br>E<br>C<br>T<br>E<br>D | Note: Some UaPs are not AEs. Report these events via an ORIO. Submit AE/ORIO report within 14 calendar days of becoming aware of event. Assess SAE to determine if UaP (see below for UaP criteria). Non-Serious Adverse Event Report in aggregate form via AE/ORIO report in conjunction with completion of the SCR. Assess AE to determine if UaP (see below for UaP criteria). | Serious Adverse Event <sup>2</sup> Report in aggregate form via separate AE/ORIO submission in conjunction with SCR. Non-Serious Adverse Event -Do not report to IRB- Study teams should continue to monitor and log events as they occur for sponsor reporting purposes. |
| E | Serious Adverse Event <sup>1</sup> , <sup>2</sup> Submit AE/ORIO report within 14 calendar days of becoming aware of event. | For ALL Unrelated & Expected Adverse Events -Do not report to IRB- |
| PECT | Non-Serious Adverse Event (Moderate/Grade 2*) -Do not report to IRB- Study teams should continue to monitor and log events as they occur. If any events appear to be occurring at a frequency greater than previously known or expected, report as unexpected within 14 calendar days of identifying trend. | Study teams should continue to monitor and log events as they occur. If any events appear to be occurring at a severity or frequency greater than previously known or expected, report as 'unexpected' per |
| E<br>D | Non-Serious Adverse Event (Mild/Grade 1*) -Do not report to IRB- Study teams should continue to monitor and log events as they occur. If any events appear to be occurring at a frequency greater than previously known or expected, report as unexpected within 14 calendar days of identifying trend. | these guidelines within 14 calendar days of identifying this trend. |

#### 1.1.4 Serious Adverse Event Reporting

We will report serious adverse events according to the Office of Research timetable above. DSC described in section 8.2. We do not anticipate any study-related serious adverse events to occur as this is a study with no more than minimal risk.

#### 1.1.5 Reporting Events to Participants

Not applicable – Any adverse events that may happen will likely be due to individual differences, e.g. baseline mental and physical health status, instead of systemic issues.

# 1.1.6 Reporting of Pregnancy

N/A

#### 1.2 Unanticipated Problems

#### 1.2.1 Definition of Unanticipated Problems (UP)

The Office for Human Research Protections (OHRP) considers unanticipated problems involving risks to participants or others to include, in general, any incident, experience, or outcome that meets <u>all</u> of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are
  described in the protocol-related documents, such as the Institutional Review Board (IRB)approved research protocol and informed consent document; and (b) the characteristics of the
  participant population being studied;
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

## 1.2.2 Unanticipated Problem Reporting

According to UM Medical School Office of Research guidelines:

Serious unanticipated problems and Unanticipated Adverse Device Effects (UADEs) must be reported within 7 calendar days of the problem (or within 7 calendar days of the study team becoming aware of the problem). Non-serious unanticipated problems must be reported within 14 calendar days of the problem (or within 14 calendar days of the study team becoming aware of the problem).

If the unanticipated problem involved one or more persons experiencing actual harm, report the unanticipated problem as an adverse event. Refer to the AE Reporting page (https://az.research.umich.edu/medschool/guidance/adverse-event-reporting) and follow the instructions provided, using the external or internal form as appropriate.

If a person did not experience actual harm but an unanticipated problem entailed potential harm, and/or risk of harm to subjects or others, refer to the ORIO Reporting page (https://az.research.umich.edu/medschool/guidance/other-reportable-information-or-occurrence-orio) and follow the instructions provided.

If the IRB concurs that an event is an unanticipated problem the study team will follow the policies and procedures outlined in the University of Michigan Human Research Protection Plan Operations Manual, part 12.

# 1.2.3 Reporting Unanticipated Problems to Participants

N/A

#### **2 STATISTICAL CONSIDERATIONS**

### 2.1 Study Hypotheses

To increase the uptake of COVID-19 vaccinations amongst African American/Black and Latinx persons living in the counties of Washtenaw, Kent, Wayne, and Genesee.

1: Increase understanding of the barriers and drivers of vaccine uptake and hesitancy;
2: Increase vaccine uptake and decrease vaccine hesitancy through the implementation and evaluation of a multilevel intervention; and maintain, enhance, and evaluate the effectiveness of the CIVIC partnership to equitably engage all partners.

#### 2.2 Sample Size Determination

PIs Resnicow and Spino have calculated sample size to account for power and individually randomized control trial.

# 2.3 Populations for Analyses

Individuals enrolled in the study will be from predominately African American/Black and Latinx populations.

#### 2.4 Statistical Analyses

#### 2.4.1 General Approach

We will follow international guidelines for analysis and reporting of individually randomized clinical trials. We will first examine the distributions of all study variables to assess missing data, possible coding errors, and distributional form, including skewness, variance, and extreme values.

Participants will see a public "control" website until their group changes into Intervention.

\*\*While the enrollment period is open throughout the intervention, only those who complete the baseline prior to the first bi-monthly check-in will have a tailored text message experience.

## 2.4.2 Analysis of the Primary Efficacy Endpoint(s)

For the primary outcome (vaccine uptake), All data will be de-identified to ensure confidentiality of participants, with results presented in summary to protect confidentiality. Analysis of quantitative questionnaire data will involve descriptive statistics, comparison of years 1-5, and examination by partner role (community or academic). Given the small number of SC members (n=19), statistical tests of significance will not be used; rather, we will identify trends for further discussion. We will use a systematic process of coding and constant comparison of all qualitative data to conceptualize group content<sub>127</sub> and to consider similarities and differences in responses for different groups (e.g., academic, community). Key quotes from the qualitative data will be selected to illustrate themes.

Descriptive statistics will be tabulated and graphical methods will be used to characterize individuals and churches. In Aim 2, summaries over time also provides information on intervention status to allow consideration of selection biases and balance. An intention-to-treat approach will be used to define the

analysis population: all participants enrolled in each randomized church for Aim 2 will be analyzed. We will summarize the extent of missing data over time for the primary endpoints. Differences in participant demographics and baseline characteristics between those with and without missing follow-up data will be given overall and by intervention group. Two-sided p-value will be reported and no adjustments for multiplicity will be made. Thus, p-values for secondary and exploratory outcomes will be interpreted with caution. Confidence intervals will be provided to summarize differences between interventions. A statistical analysis plan will be finalized prior to locking the databases. The primary outcome is the binary variable of patient reported vaccine uptake over the 6 month assessment period of the stepped wedge. Analyses will use a generalized linear mixed model with a logit link to account for the binary primary outcome; vaccinated (YES/NO). The model addresses the stepped-wedge design features including adjusting for calendar time as a fixed effect (time period) and an indicator variable that describes the treatment in each cluster (church) at each time. Given the cluster randomized nature and cohort followup in our stepped-wedge design, we will include a random intercept to account for church clustering (ICC) and a random effect for individuals in the model. An exchangeable correlation matrix that assumes similar correlation between outcomes for participants within the same church will be used. The primary statistic of interest is in the odds of vaccination between the intervention and waiting conditions, controlling for church level clustering (ICC) as well as individual level covariates, e.g., age, gender, income, education, all of which have been shown to influence vaccine uptake. Relationships between the demographics and outcome variables will be examined in bivariate analyses (Pearson and Spearman correlations, t-tests, and x2-tests). The selection of appropriate covariates for multivariable analyses will follow the variable selection approach of Heinze et al<sub>15,16</sub> that incorporates background knowledge as well as statistical criteria (such as significance of covariates with p < 0.05 or Akaike information criterion). Continuous variables such as our secondary outcome, i.e., intentions to vaccinate, will be analyzed similarly, using the identity link and the normal distribution. A priori interaction terms (intervention effect modifiers) that will be test include gender, income, education, church denomination, and ethnic identity. We will also test time interactions with treatment condition. This will allow us to determine if different lengths of exposure to the intervention yield greater outcomes, i.e., dose response effects. We expect missingness of vaccine data to be modest (< 20%), and our models account for any missingness at random. If there is substantial missingness or missingness not at random, we will use the most advanced missing data handling methods (e.g., multiple group multiple imputation) to maintain sample size and methods such as selection and pattern mixture modeling 17. Sensitivity analyses for each Aim's primary endpoint will be performed to assess the impact of missingness assumptions and approach on study conclusions.

#### Mediation Analyses.

We will use mediation analyses 18 19,20-22 under the direction of Drs. Resnicow and Spino to examine whether intervention effects on vaccine uptake and vaccine intentions, if observed, can be explained by changes in key psychosocial variables. Similar analyses will be conducted for the Aim 2 study. Specifically, we will examine whether changes in intervention targets such as vaccine attitudes, vaccine barriers, vaccine confidence, autonomous motivation, social norms, etc. account for intervention effects. Full mediation, a rare phenomenon, occurs when the association between treatment and outcome is fully eliminated in regression analyses. Mediation will be tested in a three-step process.21 First, the mediator must be affected by the independent variable (IV) of intervention. Second, the intervention must be shown to affect outcomes. Finally, it must be shown that when the dependent variable is regressed on both the independent and mediator(s), the association between IV and outcomes is attenuated. We will estimate the direct and indirect effects of the mediating variables on primary outcomes and the structural relationships (or paths) linking them using the causal inference approaches to measure the direct and effects22-24. In addition to the regression approach, we will also

use structural equation modeling (SEM) to test and visualize mediation effects. We will examine the mediators using the R package lavaan to determine indirect effects using bootstrapping. Bootstrapping does not assume normality of the product term used to examine indirect effects. Moreover, lavaan can use full information maximum likelihood estimation to efficiently address any missing data that is either missing completely at random or missing at random in any of these constructs. Finally, we will explore whether improvements in primary outcomes are associated with different exposures such as time in the social marketing intervention or number of Champion contacts.

## 2.4.3 Analysis of the Secondary Endpoint(s)

Vaccine intentions will be assessed by asking, on a scale of 0-10, "how likely is it that you will get the COVID-19 vaccine?", with 0 being very unlikely and 10 being very likely. This will be analyzed using linear regression as described in the data analysis section. "

# 2.4.4 Safety and Interim Analyses

Safety monitoring, classification of events and reporting are described in section 8. While there are no planned interim analyses other than what is done for study data safety along enrollment for the study, we may begin analysis sooner.

- The DSC members will review the following on an ongoing basis. Number screened, number enrolled, number withdrawn.
- Demographics for patients enrolled in control and intervention clinics.
- Adverse events analysis which will include descriptive analyses of the adverse event, severity, whether unexpected or expected, whether or not there were associated hospitalizations.

#### 2.4.5 Baseline Descriptive Statistics

#### 2.4.6 Tabulation of Individual Participant Data

Individual participant data will not be listed by measure and time point except for safety monitoring and reporting to IRB— and then only as aggregate and not identifiable, as outlined in section 8.

#### 2.4.7 Exploratory Analyses

### 3 SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 3.1 Regulatory, Ethical, and Study Oversight Considerations

#### 3.1.1 Informed Consent Process

This study protocol will not be implemented until reviewed and approved by the University of Michigan IRB. Potential subjects who approach study staff in person, via phone, in writing or via email, will be contacted by study staff, informed about the study and presented with the option to participate. Informed consent will be obtained prior to participation by study staff. Subjects will be informed in all cases about their rights as research subjects. Their participation is voluntary. They may decline participation without penalty or loss of any healthcare benefit or service to which they are entitled. All recruiting site personnel convey this information through the written and verbal consent process.

# 3.1.1.1 Consent/assent and Other Informational Documents Provided to participants

Consent will be obtained through the study website. Instead of a signature, they will be asked if they agree to be in the study. Answering "yes" to that question indicates consent to enroll in the study. The consent form describes in detail the study intervention, study procedures, risks and benefits, and contact information for the study team. Copy of the consent forms (one for patients enrolled to serve as controls and other for patients enrolled to receive intervention) are uploaded in eResearch.

#### 3.1.1.2 Consent Procedures and Documentation

Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. The consent process will be completed electronically through the study website.

The participant will sign/say yes to and complete the informed consent process prior to any procedures being done specifically for this study and activities that are not unregulated. Participants will be informed that participation is voluntary and that they may withdraw from the study at any time, without negative impact to them (without prejudice). An electronic copy of the informed consent document will be given or sent to the participants for their records. The informed consent process will be conducted and documented in the source document (including the date), and the form signed, before the participant undergoes any study-specific procedures. The rights and welfare of the participants will be emphasized and consent will include a specific statement that the quality of their medical care will not be adversely affected if they decline to participate in this study.

#### 3.1.2 Study Discontinuation and Closure

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigator, funding agency, and regulatory authorities as appropriate. If the study is prematurely terminated or suspended, the Principal Investigator (PI) will promptly inform study participants, the Institutional Review Board (IRB), and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the sponsor, DSC and IRB.

#### 3.1.3 Confidentiality and Privacy

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their interventions. This confidentiality is extended to cover testing of biological samples, patient-reported measures (either during coaches or study surveys) and clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. In this case the clinical study site will permit access to such records.

The study participant's contact information will be securely stored on a secure server at U-M for as long a period as dictated by the reviewing IRB, institutional policies, or sponsor requirements.

The database that contains survey results and clinical data will only be identified by study ID's. A separate file will be created to link the participant's name and other identifiable data to the study ID. Only the core study team (e.g. PI and research assistants) will have access to the password protected linking file. We do not anticipate any information to be identifiable without the linking file. Only key personnel will be able to have access to identifiable information on participants.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the University of Michigan. All transferred data will abide by local and UM policies regarding sharing data and encryption. The study data entry and study management systems used by clinical sites and by University of Michigan research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the University of Michigan.

#### Certificate of Confidentiality

To further protect the privacy of study participants, a Certificate of Confidentiality will be issued by the National Institutes of Health (NIH). This certificate protects identifiable research information from forced disclosure. It allows the investigator and others who have access to research records to refuse to disclose identifying information on research participation in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level. By protecting researchers and institutions from being compelled to disclose information that would identify research participants, Certificates of Confidentiality help achieve the research objectives and promote participation in studies by helping assure confidentiality and privacy to participants.

# 3.1.4 Future Use of Stored Specimens and Data

- Deidentified data will be retained for study record keeping purposes and future research, it will be stored, indefinitely, on secure servers at U-M.
  - Data will be stripped of all identifiers before storage.

#### 3.1.5 Key Roles and Study Governance

# **Principle Investigator:**

Kenneth Resnicow, PhD,
Irwin M. Rosenstock Collegiate Professor
Associate Director, Community Outreach and Health Disparities Research Rogel Cancer Center
Department of Health Behavior Health Education
University of Michigan
Building 16, North Campus Research Complex Office 16-G036E 2800 Plymouth Rd.
Ann Arbor MI 48109
United States
kresnic@umich.edu

**Co-investigators/Study Team**: Larry An, M.D., Chris Coombe, Barbara Israel, Ph.D., Erica Marsh, M.D., M.P.H., Catherine Spino, Ph.D., Charles Williams, Charley Jiang, Emerson Delacroix, LLP, MACP, Patricia Piechowski, Arthi Ramakrishnan, Liz Bacon, MPH, Mary Beth Damm, MPP, Kirsten Trzeciak.

#### 3.1.6 Safety Oversight

Safety oversight will be under the direction of a Data and Safety Committee (DSC) composed of individuals with the appropriate expertise. The DSC will consist of selected members who have no conflicts of interest with the study. The DSC will be led by the PI. He has served on other DSCs and is both a clinical leader and well-established researcher. As needed, the PI and study biostatistician will be available to provide input and attend the DSC meetings. The DSC has approved initiation of the proposed study for enrollment of human subjects, evaluate the progress of the study at initiation, when enrollment is 25% complete, 50% complete, and 100% complete. Additionally, if the study is slow to recruit, the DSC will meet at least yearly. In addition, urgent or emergent meetings of the DSC may be called at any time by the chair of the DSC or NIH project officer in event of any issues regarding patient safety. At this time, each data element that the DSC needs to assess will be clearly defined. DSC reports will be included in status reports (RPPR reporting) to the NIH yearly.

#### 3.1.7 Clinical Monitoring

N/a

# 3.1.8 Quality Assurance and Quality Control

To ensure consistent delivery of the intervention and uniform application of enrollment and data collection protocols, we hosted a kick-off meeting in Year 1 attended by prospective Religious and Spiritual Leaders, research staff, project support and Steering Committee members. Goals of the study were discussed along with design and procedures. Study team members have been split into teams and assigned aspects of the study to develop and give input on study materials development. In addition, we brought in experts in quality improvement (through UM Quality and Innovation Program) and leaders on the study team in continuous quality improvement (CQI). With study team member input, we have developed a study team communication plan for study personnel, staff, co-investigators, as well as providers and staff in involved clinics. We are working with staff at UM to develop an online project website, and there will be an additional secure/password protected feature for providers from involved clinics to sign in and learn more about the study. Descriptions of the study will be produced in a variety of formats for distribution via group emails and as handouts in the community that include study key facts for consistency.

In addition, for specific study procedures, we will produce data collection manuals with detailed instructions for issues such as how to note missing data, how to make changes on data collection forms, and how to adjudicate decisions when survey response options are unclear and have this reviewed by our colleague experts in CQI. In addition, once enrollment begins, data quality issues will be discussed at weekly meetings between project staff and the PI. Data integrity and completeness will be checked periodically by research personnel and reported at biweekly team meetings as described previously in section 8.2.

Quality control (QC) procedures will be implemented beginning with the data entry systems and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to staff for clarification/resolution.

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

Rigor and reproducibility will be maximized by quality control of all study protocols and procedures and by using a robust experimental design for the intervention. This study applies high standards in its methodology and its analysis plan which will be continued through interpretation and results reporting. We will be transparent in reporting experimental details so that others may reproduce and extend the findings in the future.

#### 3.1.9 Data Handling and Record Keeping

Data will be deidentified for indefinite storage on secured servers at U-M, to assist with future research. Study data will be stored in a relational database on a separate highly restricted secure server. Databases will be backed up daily to an offsite NAS storage device using automatic backup software that is available 24/7 except for scheduled maintenance. Only the primary investigators and other authorized research team members named in this application will have access to the de-identified data. These standards will help ensure that violations of confidentiality will be minimal.

# 3.1.9.1 Data Collection and Management Responsibilities

All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Study data will be stored on research compliant servers provided by the University of Michigan. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

#### 3.1.9.2 Study Records Retention

Study documents will be retained until the formal discontinuation of the study intervention. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained.

#### 3.1.10 Protocol Deviations

It is the responsibility of the PI to use continuous vigilance to identify and report deviations. All deviations will be addressed in study source documents, reported to the NIH Program Official and University of Michigan Institutional Review Board (IRB). The site investigator is responsible for knowing and adhering to the reviewing IRB requirements.

# 3.1.11 Publication and Data Sharing Policy

This study will be conducted in accordance with the following publication and data sharing policies and regulations:

National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive <a href="PubMed Central">PubMed Central</a> upon acceptance for publication.

This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers years after the completion of the primary endpoint by contacting Ken Resnicow, Ph.D.

#### 3.1.12 Conflict of Interest Policy

The independence of this study from any actual or perceived influence is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. The study leadership in conjunction with the NIH and U-M that have established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

# 3.2 Additional Considerations

Not applicable.

#### 3.3 Abbreviations

| AA | African Americans |
|-------|------------------------------------------------------------------|
| AE | Adverse Event |
| CIVIC | Community-centered Interventions for Vaccine Uptake for COVID-1( |
| DSC | Data Safety Committee |
| GCP | Good Clinical Practice |
| G2YMI | Getting to Yes, Michigan! |
| HIPAA | Health Insurance Portability and Accountability Act |
| IRB | Institutional Review Board |
| LX | Latinx |
| NCT | National Clinical Trial |
| NIH | National Institutes of Health |
| PI | Principal Investigator |
| RA | Research assistant / research associate |
| U-M | University of Michigan |
| UP | Unanticipated Problem |
| US | United States |

#### 3.4 Protocol Amendment History

# Amendment #1: Ame00123018 Recruitment

- 1. Recruitment materials have been updated to exclude outdated language not approved in original app. These added recruitment materials for use at churches (e.g. posters, business cards, prompts for written communications from RSL to church attendees).
- 2. Additional churches have opted to participate and added to Participating sites.
- 3. Spanish consent has additional sentence added.
- 4. Updated study email from gettingtoyesmichigan@umich.edu to gettingtoyesmi@med.umich.edu.

## Amendment #2: Ame00123968 Staff, Church Recruitment Pkt/Flyers

- 1. Study Team Members have been updated to include new RAs and remove staff off the project.
- 2. Updated church fliers and welcome packet to include HUM# and reformatted for improved aesthetic.
- 3. Fully executed Collaborating Institution and Project Participation Agreements added to each church in 3-1.1\* Performance Sites.
- 4. Removed churches from section 3-1.1 Performance Sites that are no longer participating in the study.

#### Amendment #3: Ame00128520 RCT

- 1. Changed statistical design from Stepped Wedge to RCT
- 2. Changed eligibility criteria to include updated booster guidelines per CDC
- 3. Expanded recruitment to include non-church community members to allow for public recruitment events, rather than faith-based recruitment events
- 4. Recruiting Vaccine Champions who will go through virtual training only. Newly recruited Vaccine Champions will not receive incentives and will not interact directly with participants.
- 5. Updated consent to include eligibility and recruitment changes noted above.

- 6. Updated enrollment numbers
- 7. Included of MMS messages
- 8. Update study team members.

#### Amendment #4: Ame00133699 Audit Edits

- 1. Add completed GCP trainings for all study team members.
- 2. Update Protocol
- 3. Update funding
- 4. Update consent
- 5. Update DSMB to DSC

#### Amendment # 5: Ame00136269 SPAN-flyer

- 1. Add Spanish translation of approved English recruitment flyer.
- 2. Edit team members.

#### Amendment #6: Ame00137511 New Ads, Staff

- 1. Add new social media ads
- 2. Edit team members

#### Amendment-7: Ame00138260 Data Direct, Staff

- 1. Recruitment Expansion to add Data Direct added to Protocol and application. Added recruitment Scripts in English and Spanish to 08-1.
  - 2. Edit team members

#### Amendment-8: Ame00141536 Omicron Booster

- 1. Survey and content will be updated to reflect the FDA updated guidelines for defining "up-to-date" as receiving the bivalent ("Omicron") booster.
  - 2. Staff members added/removed.
  - 3. Enrollment target is increased to 800 to have power for analysis after guide changes.

#### Amendment-9: Ame00144824 Update Articulate, Enrollment

- 1. Increase Enrollment to 1000 to increase population eligible for analysis.
- 2. Update Vaccine Champion Articulate Training with up-to-date content related to Sept 2023 vaccine.
  - 3. Update Public Articulate Training with up-to-date content related to Sept 2023 vaccine.

#### Amendment-10: Ame00146052 Protocol

1. Update protocol.

# 3.5 Appendices

# APPENDIX 1: OUTCOME MEASURES

| Variable | Time point(s) | Variable | Outcome type |
|---|---|---|---|
| | | type | |
| Demographics/patient characteristics (age, sex, gender, race, ethnicity, | t(0) | continuous, | N/A |
| education, income) | | categorical | |
| Participant SMS/MMS responses response for vaccine uptake | | continuous, | primary |
| | | categorical | |
| Participant perceptions | t(1), t(2), t(3) | continuous | exploratory |
| Vaccine intention | t(1), t(2), t(3) | continuous | exploratory |

#### 4 REFERENCES

- 1. Brown EJ, Polsky D, Barbu CM, Seymour JW, Grande D. Racial Disparities In Geographic Access To Primary Care In Philadelphia. Health Aff (Millwood). 2016;35(8):1374-1381.
- 2. Mahmoudi E, Jensen GA. Diverging racial and ethnic disparities in access to physician care: comparing 2000 and 2007. Med Care. 2012;50(4):327-334.
- 3. Grobman WA, Bailit JL, Rice MM, et al. Racial and ethnic disparities in maternal morbidity and obstetric care. Obstet Gynecol. 2015;125(6):1460-1467.
  - 4. Webb Hooper M, Napoles AM, Perez-Stable EJ. COVID-19 and Racial/Ethnic Disparities. JAMA. 2020;323(24):2466-2467.
- 5. Kulwicki AD, Miller J, Schim SM. Collaborative partnership for culture care: enhancing health services for the Arab community. J Transcult Nurs. 2000;11(1):31-39.
  - 6. Agency for Healthcare Research and Quality. National Healthcare Quality and Disparities Reports.
- http://www.ahrq.gov/research/findings/nhqrdr/index.html. Accessed January 31, 2021.
- 7. Laurencin CT, McClinton A. The COVID-19 Pandemic: a Call to Action to Identify and Address Racial and Ethnic Disparities. J Racial Ethn Health Disparities. 2020;7(3):398-402.
  - 8. Dorn AV, Cooney RE, Sabin ML. COVID-19 exacerbating inequalities in the US. Lancet. 2020;395(10232):1243-1244.
  - 9. Yancy CW. COVID-19 and African Americans. JAMA. 2020;323(19):1891-1892.
- 10. State of Michigan. Coronavirus: Michigan Data. 2021; https://www.michigan.gov/coronavirus/0,9753,7-406-98163\_98173---,00.html. Accessed January 31, 2021.
- 11. State of Michigan. Governor Whitmer Signs Executive Order Creating the Michigan Coronavirus Task Force on Racial Disparities. 2020; https://www.michigan.gov/whitmer/0,9309,7-387-90499-526478--
- ,00.html#:~:text=The%20task%20force%20will%20investigate,physical%20and%20mental%20health%20care. Accessed January 31, 2021.
- 12. Michigan Department of Health & Human Services. Michigan Coronavirus Racial Disparities Task Force: Interim Report. 2020; https://content.govdelivery.com/attachments/MIEOG/2020/12/03/file\_attachments/1616552/COVID-19%20Task%20Force%20on%20Racial%20Disparities%20Interim%20Report.pdf. Accessed January 31, 2021.
- 13. Centers for Disease Control and Prevention. COVID-19 Vaccinations in the United States. 2021; https://covid.cdc.gov/covid-data-tracker/#vaccinations. Accessed January 31, 2021.
- 14. State of Michigan. COVID-19 Vaccine Dashboard. 2021; https://www.michigan.gov/coronavirus/0,9753,7-406-98178\_103214-547150--,00.html. Accessed January 31, 2021.
- 15. Michigan Department of Health & Human Services. Racial Disparity Task Force January 22, 2021. 2021; https://www.michigan.gov/documents/mdhhs/Racial\_Disparities\_Task\_Force\_714385\_7.pdf. Accessed January 31, 2021.
- 16. U.S. Census Bureau. QuickFacts: Genessee County, Michigan. 2019; https://www.census.gov/quickfacts/fact/table/geneseecountymichigan/PST045219. Accessed January 31, 2021.

- 17. U.S. Census Bureau. QuickFacts: Kent County, Michigan. 2019;
- https://www.census.gov/quickfacts/fact/table/kentcountymichigan/PST045219. Accessed January 31, 2021.
  - 18. U.S. Census Bureau. QuickFacts: Washtenaw County, Michigan. 2019;
- https://www.census.gov/quickfacts/fact/table/washtenawcountymichigan/PST045219. Accessed January 31, 2021.
  - 19. U.S. Census Bureau. QuickFacts: Wayne County, Michigan. 2019;
- https://www.census.gov/quickfacts/fact/table/waynecountymichigan/PST045219. Accessed January 31, 2021.
  - 20. Charter County of Wayne Michigan. Wayne County COVID-19 Dashboard. 2021;
- https://wayne.maps.arcgis.com/apps/opsdashboard/index.html#/d04fff4645b140319fad972eb3740550. Accessed January 31, 2021.
- 21. University of Michigan Office of the Vice President for Communications. Majority of Detroiters say they're unlikely to get COVID-19 vaccine, U-M survey says. 2020; https://news.umich.edu/majority-of-detroiters-say-theyre-unlikely-to-get-covid-19-vaccine-u-m-survey-says/. Accessed January 31, 2021.
- 22. Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202.
- 23. Israel BA, Schulz AJ, Parker EA, et al. Critical Issues in Developing and Following CBPR Principles. In: Wallerstein N, Duran B, Oetzel JG, Minkler M, eds. Community-Based Participatory Research for Health: Advancing Social and Health Equity. 3rd ed. Hoboken, NJ: Jossey-Bass; 2018:31-46.
- 24. Schulz AJ, Mehdipanah R, Chatters LM, Reyes AG, Neblett EW, Jr., Israel BA. Moving Health Education and Behavior Upstream: Lessons From COVID-19 for Addressing Structural Drivers of Health Inequities. Health Educ Behav.. 2020;47(4):519-524.
- 25. Braveman P, Egerter S, Robert Wood Johnson Foundation Commission to Build a Healthier America. Overcoming Obstacles to Health in 2013 and Beyond. 2013; https://www.rwjf.org/en/library/research/2013/06/overcoming-obstacles-to-health-in-2013-and-beyond.html. Accessed January 31, 2021.
- 26. Cacari-Stone L, Wallerstein N, Garcia AP, Minkler M. The promise of community-based participatory research for health equity: a conceptual model for bridging evidence with policy. Am J Public Health. 2014;104(9):1615-1623.
- 27. Wallerstein N, Duran B. Theoretical, Historical, and Practice Roots of CBPR. In: Wallerstein N, Duran B, Oetzel JG, Minkler M, eds. Community-Based Participatory Research for Health: Advancing Social and Health Equity. 3rd ed. Hoboken, NJ: Jossey-Bass; 2018:17-30.
- 28. Israel BA, Schulz AJ, Coombe CM, et al. Community-Based Participatory Research: An Approach to Research in the Urban Context. In: Galea S, Ettman CK, Vlahov D, eds. Urban Health. New York, NY: Oxford University Press; 2019.
- 29. Ward M, Schulz AJ, Israel BA, Rice K, Martenies SE, Markarian E. A conceptual framework for evaluating health equity promotion within community-based participatory research partnerships. Eval Program Plann. 2018;70:25-34.
- 30. Resnicow K, Coleman-Wallace D, Jackson A, et al. Dietary Change through Black Churches: Baseline Results and Program Description of the Eat for Life Trial. J Cancer Educ.. 2000;15:156-163.
- 31. Resnicow K, Taylor R, Baskin M. Results of Go Girls: A nutrition and physical activity intervention for overweight African American adolescent females conducted through Black churches. Obes Res. 2005;13(10):1739-1748.

- 32. Resnicow K, Campbell MK, Carr C, et al. Body and soul. A dietary intervention conducted through African-American churches. Am J Prev Med. 2004;27(2):97-105.
- 33. Resnicow K, Wallace DC, Jackson A, et al. Dietary change through African American churches: baseline results and program description of the eat for life trial. J Cancer Educ. 2000;15(3):156-163.
- 34. Resnicow K, Jackson A, Wang T, et al. A motivational interviewing intervention to increase fruit and vegetable intake through Black churches: results of the Eat for Life trial. Am J Public Health. 2001;91(10):1686-1693.
- 35. Resnicow K, Jackson A, Braithwaite R, et al. Healthy Body/Healthy Spirit: a church-based nutrition and physical activity intervention. Health Educ Res. 2002;17(5):562-573.
- 36. Campbell MK, Resnicow K, Carr C, Wang T, Williams A. Process evaluation of an effective church-based diet intervention: Body & Soul. Health Educ Behav.. 2007;34(6):864-880.
- 37. Allicock M, Johnson LS, Leone L, et al. Promoting fruit and vegetable consumption among members of black churches, michigan and north Carolina, 2008-2010. Prev Chronic Dis. 2013;10:E33.
- 38. Langford AT, Resnicow K, Beasley DD. Outcomes from the Body & Soul Clinical Trials Project: a university-church partnership to improve African American enrollment in a clinical trial registry. Patient Educ Couns. 2015;98(2):245-250.
- 39. Berkley-Patton J, Bowe Thompson C, Goggin K, et al. A religiously-tailored, multilevel intervention in African American churches to increase HIV testing: Rationale and design of the Taking It to the Pews cluster randomized trial. Contemp Clin Trials. 2019;86:105848.
- 40. Resnicow K, Davis RE, Zhang G, et al. Tailoring a fruit and vegetable intervention on novel motivational constructs: results of a randomized study. Ann Behav Med. 2008;35(2):159-169.
- 41. Resnicow K, Zhou Y, Hawley S, et al. Communication preference moderates the effect of a tailored intervention to increase colorectal cancer screening among African Americans. Patient Educ Couns. 2014;97(3):370-375.
- 42. Woolford SJ, Clark SJ, Strecher VJ, Resnicow K. Tailored mobile phone text messages as an adjunct to obesity treatment for adolescents. J Telemed Telecare. 2010;16(8):458-461.
- 43. Wilson DK, Alia KA, Kitzman-Ulrich H, Resnicow K. A pilot study of the effects of a tailored web-based intervention on promoting fruit and vegetable intake in African American families. Child Obes. 2014;10(1):77-84.
- 44. Beebe J. Rapid Qualitative Inquiry: A Field Guide to Team-Based Assessment. Second ed. Lanham, MD: Rowman & Littlefield Publishers; 2014.
- 45. Abramowitz SA, McLean KE, McKune SL, et al. Community-centered responses to Ebola in urban Liberia: the view from below. PLoS Negl Trop Dis. 2015;9(4):e0003706.
- 46. Lee-Kwan SH, DeLuca N, Adams M, et al. Support services for survivors of ebola virus disease Sierra Leone, 2014. MMWR Morb Mortal Wkly Rep. 2014;63(50):1205-1206.
- 47. Summers A, Nyenswah TG, Montgomery JM, et al. Challenges in responding to the ebola epidemic four rural counties, Liberia, August-November 2014. MMWR Morb Mortal Wkly Rep. 2014;63(50):1202-1204.
- 48. Neal JW, Neal ZP, VanDyke E, Kornbluh M. Expediting the Analysis of Qualitative Data in Evaluation: A Procedure for the Rapid Identification of Themes From Audio Recordings (RITA). Am J Eval. 2015;36(1):115-132.

- 49. Guest G, MacQueen KM, Namey EE. Applied Thematic Analysis. Thousand Oaks, CA: SAGE Publications; 2011.
- 50. Bhattacharya K. Fundamentals of qualitative research: A practical guide. New York, NY: Routledge; 2017.
- 51. Oganesyan N. Positive COVID-19 Messaging on TV Can Persuade Resistant Viewers, The Protector Coalition Says. 2021; https://variety.com/2021/tv/news/positive-tv-messaging-coronavirus-the-protector-coalition-1234885193/. Accessed February 1, 2021.
- 52. Baskin M, Resnicow K, Campbell M. Conducting Health Interventions in Black Churches: A Model for Building Effective Partnerships. Ethnic Dis.. 2001;11:823-833.
- 53. Andrews AM, Zhang N, Magee JC, Chapman R, Langford A, Resnicow k. Increasing donor designation through black churches: results of a randomized trial. Prog Transplant.. 2012;22(161-167).
- 54. Fuemmeler BF, Masse LC, Yaroch AL, et al. Psychosocial mediation of fruit and vegetable consumption in the Body and Soul effectiveness trial. Health Psychology. 2006;25(4):474-483.
- 55. Allicock M, Campbell MK, Valle CG, Carr C, Resnicow K, Gizlice Z. Evaluating the Dissemination of Body & Soul, an Evidence-based Fruit and Vegetable Intake Intervention: Challenges for Dissemination and Implementation Research. J Nutr Educ Behav. 2012;44(6):530-8.
- 56. Cassel KD, Braun K, Ka'opua L, Soa F, Nigg C. Samoan body and soul: adapting an evidence-based obesity and cancer prevention program. Qual Health Res. 2014;24(12):1658-1672.
- 57. Catley D, Puoane T, Goggin K, et al. Adapting the Diabetes Prevention Program for low- and middle-income countries: preliminary implementation findings from lifestyle Africa. Transl Behav Med. 2020;10(1):46-54.
- 58. do Valle Nascimento TMR, Resnicow K, Nery M, et al. A pilot study of a Community Health Agent-led type 2 diabetes self-management program using Motivational Interviewing-based approaches in a public primary care center in São Paulo, Brazil. BMC Health Serv Res. 2017;17(1):32.
- 59. McMaster F, Resnicow K. Validation of the one pass measure for motivational interviewing competence. Patient Educ Couns. 2015;98(4):499-505.
- 60. Hemming K, Girling A. A menu-driven facility for power and detectable-difference calculations in stepped-wedge cluster-randomized trials. Stata Journal. 2014;14(2):363-380.
  - 61. Kaiser Family Foundation. KFF Health Tracking Poll/ KFF COVID-19 Vaccine Monitor: December 2020 Washington, D.C. 2020.
- 62. Pew Research Center. Intent to Get a COVID-19 Vaccine Rises to 60% as Confidence in Research and Development Process Increases. 2020.
- 63. Murray DM. Intraclass correlation among measures related to alcohol use by school aged adolescents: estimates, correlates and applications in intervention studies. J Drug Educ. 1996;26(3):207-230.
- 64. Murray DM, Alfano CM, Zbikowski SM, Padgett LS, Robinson LA, Klesges R. Intraclass correlation among measures related to cigarette use by adolescents: estimates from an urban and largely African American cohort. Addictive Behaviors. 2002;27(4):509-527.
- 65. Murray DM, Blistein JL. Methods to reduce the impact of intraclass correlation in group-randomized trials. Evaluation Review. 2003;27(1):79-103.
- 66. Resnicow K, Zhang N, Vaughan RD, Reddy SP, James S, Murray DM. When Intraclass Correlation Coefficients Go Awry: A Case Study From a School-Based Smoking Prevention Study in South Africa. Am J Public Health. 2010.

- 67. Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. Psychological Bulletin. 2007;133(4):673-693.
- 68. Hawkins R, Kreuter M, Resnicow K, Fishbein M, Dijkstra A. Understanding Tailoring in Communicating About Health. Health Educ Res. 2008;23(3):454-466.
- 69. Scheffers-van Schayck T, Mujcic A, Otten R, Engels R, Kleinjan M. The Effectiveness of Smoking Cessation Interventions Tailored to Smoking Parents of Children Aged 0-18 Years: A Meta-Analysis. Eur Addict Res. 2020:1-16.
- 70. Lustria ML, Noar SM, Cortese J, Van Stee SK, Glueckauf RL, Lee J. A meta-analysis of web-delivered tailored health behavior change interventions. J Health Commun. 2013;18(9):1039-1069.
- 71. van Keulen HM, Mesters I, Ausems M, et al. Tailored print communication and telephone motivational interviewing are equally successful in improving multiple lifestyle behaviors in a randomized controlled trial. Ann Behav Med. 2011;41(1):104-118.
- 72. Resnicow K, Davis RE, Zhang G, et al. Tailoring a fruit and vegetable intervention on novel motivational constructs: results of a randomized study. Ann Behav Med. 2008;35(2):159-169.
- 73. Bangor A, Kortum PT, Miller JT. An Empirical Evaluation of the System Usability Scale. International Journal of Human–Computer Interaction. 2008;24(6):574-594.
- 74. Williams GC, Rodin GC, Ryan RM, Grolnick WS, Deci EL. Autonomous regulation and long-term medication adherence in adult outpatients. Health Psychol. 1998;17(3):269-276.
  - 75. Williams GC, Gagne M, Ryan RM, Deci EL. Facilitating autonomous motivation for smoking cessation. Health Psychol. 2002;21(1):40-50.
- 76. Markland D, Ryan RM, Tobin VJ, Rollnick S. Motivational Interviewing and Self-Determination Theory. J Soc Clin Psychol. 2005;24(6):811-831.
  - 77. Deci E, Ryan R. Intrinsic motivation and self-determination in human behavior. New York: Plenum; 1985.
- 78. Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000;55(1):68-78.
- 79. Williams GC, Freedman ZR, Deci EL. Supporting autonomy to motivate patients with diabetes for glucose control. Diabetes Care. 1998;21(10):1644-1651.
- 80. Dempsey A, Kwan BM, Wagner NM, et al. A Values-Tailored Web-Based Intervention for New Mothers to Increase Infant Vaccine Uptake: Development and Qualitative Study. J Med Internet Res. 2020;22(3):e15800.
- 81. Belgrave FZ, Cherry VR, Cunningham D, Walwyn S, Letkala-Rennert K, Phillips F. The influence of Africentric values, self-esteem, and Black identity on drug attitudes among African American fifth graders: A preliminary study. Special Section: Africentric values, racial identity, and acculturation: Measurement, socialization, and consequences. J Black Psychol. 1994;20(2):143-156.
  - 82. Helms JE. Black and White racial identity: Theory, research, and practice. Greenwood Press. 1990;262.
- 83. Parham T, Helms J. The influence of Black students' racial identity attitudes on preferences for counselor's race. J Couns Psychol. 1981;28(3):250-257.
- 84. Resnicow K, Soler R, Braithwaite R, Selassie M, Smith M. Development and Validation of a Racial Identity Scale for African American Adolescents: The Survey of Black Life. J Couns Psychol. 1999;25(2):171-188.

- 85. Sellers RM. A call to arms for researchers studying racial identity. Special Section: Racial identity revisited. J Couns Psychol. 1993;19(3):327-332.
- 86. Resnicow K, Davis R, Zhang N, et al. Tailoring a fruit and vegetable intervention on ethnic identity: Results of a randomized study. Health Psychol. 2009;28(4):394-403.
- 87. Nicholson RA, Kreuter MW, Lapka C, et al. Unintended effects of emphasizing disparities in cancer communication to African-Americans. Cancer Epidemiol Biomarkers Prev. 2008;17(11):2946-2953.
- 88. Davis RE, Alexander G, Calvi J, et al. A new audience segmentation tool for African Americans: the black identity classification scale. J Health Commun. 2010;15(5):532-554.
- 89. Sellers RM, Rowley SA, Chavous TM, Shelton J, Smith MA. Multidimensional Inventory of Black Identity: A preliminary investigation of reliability and constuct validity. J Pers Soc Psychol. 1997;73(4):805-815.
- 90. Grobe JE, Goggin K, Harris KJ, Richter KP, Resnicow K, Catley D. Race moderates the effects of Motivational Interviewing on smoking cessation induction. Patient Educ Couns. 2020;103(2):350-358.
- 91. U.S. Department of Health & Human Services. NIH Public Health Emergency and Disaster Research Response (DR2). 2021; https://dr2.nlm.nih.gov/. Accessed February 1, 2021.
- 92. An L, Hawley S, Van Horn ML, Bacon E, Yang P, Resnicow K. Development of a coronavirus social distance attitudes scale. Patient Educ Couns. 2020.
- 93. Levesque CS, Williams GC, Elliot D, Pickering MA, Bodenhamer B, Finley PJ. Validating the theoretical structure of the Treatment Self-Regulation Questionnaire (TSRQ) across three different health behaviors. Health Educ Res. 2007;22(5):691-702.
- 94. Resnicow K, Bacon E, Yang P, Hawley S, Van Horn ML, An L. Novel Predictors of Coronavirus Protective Behaviors among US adults: The role of trait reactance, conspiracy beliefs, and belief in the apocalypse. JMIR. In Press.
- 95. Dempsey AF, Wagner N, Narwaney K, et al. 'Reducing Delays In Vaccination' (REDIVAC) trial: a protocol for a randomised controlled trial of a web-based, individually tailored, educational intervention to improve timeliness of infant vaccination. BMJ Open. 2019;9(5):e027968-e027968.
- 96. Glanz JM, Wagner NM, Narwaney KJ, et al. Web-Based Tailored Messaging to Increase Vaccination: A Randomized Clinical Trial. Pediatrics. 2020;146(5):e20200669.
- 97. Wheldon CW, Kolar SK, Hernandez ND, Daley EM. Factorial Invariance and Convergent Validity of the Group-Based Medical Mistrust Scale across Gender and Ethnoracial Identity. J Health Care Poor Underserved. 2017;28(1):88-99.
- 98. Valera P, Boyas JF, Bernal C, Chiongbian VB, Chang Y, Shelton RC. A Validation of the Group-Based Medical Mistrust Scale in Formerly Incarcerated Black and Latino Men. Am J Mens Health. 2018;12(4):844-850.
- 99. Shelton RC, Winkel G, Davis SN, et al. Validation of the group-based medical mistrust scale among urban black men. J Gen Intern Med. 2010;25(6):549-555.
- 100. Thompson HS, Valdimarsdottir HB, Winkel G, Jandorf L, Redd W. The Group-Based Medical Mistrust Scale: psychometric properties and association with breast cancer screening. Prev Med. 2004;38(2):209-218.

- 101. Quinn SC, Jamison AM, An J, Hancock GR, Freimuth VS. Measuring vaccine hesitancy, confidence, trust and flu vaccine uptake: Results of a national survey of White and African American adults. Vaccine. 2019;37(9):1168-1173.
- 102. Resnicow K, Vaughan R, Royce J, Orlandi M. Process analysis of the Kick It! smoking cessation project: What worked and why? Prev Med. 1997;26:373-381.
- 103. Resnicow K, Gobat N, Naar S. Intensifying and igniting change talk in Motivational Interviewing: A theoretical and practical framework. European Health Psychologist. 2015;Vol 17(3):102-110.
- 104. Williams GC, McGregor HA, Zeldman A, Freedman ZR, Deci EL. Testing a self-determination theory process model for promoting glycemic control through diabetes self-management. Health Psychol. 2004;23(1):58-66.
- 105. Williams GC, Niemiec CP, Patrick H, et al. The importance of supporting autonomy and perceived competence in facilitating long-term tobacco abstinence. Ann Behav Med. 2009;37(3):315-324.
  - 106. Shen L, Dillard JP. Psychometric properties of the Hong psychological reactance scale. J Pers Assess. 2005;85(1):74-81.
  - 107. Jonason PK, Knowles HM. A unidimensional measure of Hong's psychological reactance scale. Psychol Rep. 2006;98(2):569-579.
- 108. Donnell AJ, Thomas A, Buboltz WC, Jr. Psychological reactance: factor structure and internal consistency of the Questionnaire for the Measurement of Psychological Reactance. J Soc Psychol. 2001;141(5):679-687.
- 109. Hong SM, Giannakopoulos E, Laing D, Williams NA. Psychological reactance: effects of age and gender. J Soc Psychol. 1994;134(2):223-228.
  - 110. Hong S, Page S. A psychological reactance scale: Development, factor structure and reliability. Psychol Rep. 1989; 64:1323–1326.
- 111. van Prooijen JW, van Vugt M. Conspiracy Theories: Evolved Functions and Psychological Mechanisms. Perspect Psychol Sci. 2018;13(6):770-788.
- 112. Freeman D, Waite F, Rosebrock L, et al. Coronavirus conspiracy beliefs, mistrust, and compliance with government guidelines in England. Psychol Med. 2020:1-13.
  - 113. Tyminski R. Apocalyptic themes in times of trouble: when young men are deeply alienated. J Anal Psychol. 2020;65(1):27-43.
  - 114. contributors W. Apocalypticism. 2020; https://en.wikipedia.org/wiki/Apocalypticism. Accessed July 14, 2020.
- 115. Centers for Disease Control and Prevention. How to Protect Yourself & Others. 2020; https://www.cdc.gov/coronavirus/2019-ncov/prevent-getting-sick/prevention.html. Accessed July 29th, 2020.
- 116. Resnicow K, Patel MR, Green M, et al. Development of an Ethnic Identity Measure for Americans of Middle Eastern and North African Descent: Initial Psychometric Properties, Sociodemographic, and Health Correlates. J Racial Ethn Health Disparities. 2020; September 24: doi: 10.1007/s40615-020-00863-y. Online ahead of print.
- 117. Resnicow K, Strecher V, Couper MP, et al. Methodologic and Design Issues in Patient-Centered e-Health Research. Am J Prev Med. 2010;38(1):98-102.
- 118. Israel BA, Lachance L, Coombe CM, et al. Measurement Approaches to Partnership Success: Theory and Methods for Measuring Success in Long-Standing Community-Based Participatory Research Partnerships. Prog Community Health Partnersh. 2020;14(1):129-140.

- 119. Israel BA, Lantz P, McGranaghan R, Guzman JR, Lichtenstein R, Rowe Z. Documentation and evaluation of community-based participatory research partnerships: The use of in-depth interviews and closed-ended questionnaires. In: Israel BA, Eng E, Schulz AJ, Parker EA, eds. Methods in Community-Based Participatory Research for Health. 2nd ed. Hoboken, NJ: Jossey-Bass; 2012:369-403.
- 120. Quinn SC, Jamison A, An J, Freimuth VS, Hancock GR, Musa D. Breaking down the monolith: Understanding flu vaccine uptake among African Americans. SSM Popul Health. 2018;4:25-36.
- 121. Israel BA, Lichtenstein R, Lantz P, et al. The Detroit Community-Academic Urban Research Center: development, implementation, and evaluation. J Public Health Manag Pract. 2001;7(5):1-19.
- 122. Schulz AJ, Israel BA, Lantz P. Instrument for evaluating dimensions of group dynamics within community-based participatory research partnerships. Eval Program Plann. 2003;26(3):249-262.
- 123. Coombe C. Participatory Approaches to Evaluating Community Organizing and Coalition Building. In: Minkler M, ed. Community Organizing and Community Building for Health and Welfare. New Brunswick, NJ: Rutgers University Press; 2012.
- 124. Cousins JB, Chouinard JA. Participatory Evaluation up Close: An Integration of Research-Based Knowledge. Charlotte, NC: Information Age Publishing; 2012.
- 125. Goold S, Rowe Z, Calhoun K, et al. The State as Community in Community-Based Participatory Research. Prog Community Health Partnersh. 2016;10(4):515-522.
  - 126. Clark VLP, Creswell JW. Designing and Conducting Mixed Methods Research. 3rd ed. Thousand Oaks, CA: SAGE Publishing; 2017.
  - 127. Charmaz K. Constructing Grounded Theory. Second ed. Thousand Oaks, CA: Sage Publications; 2014.
  - 128. Rossi PH, Freeman HE, Lipsey MW. Evaluation: A Systematic Approach. 6th ed. Thousand Oaks, CA: SAGE Publishing; 1999.
- 129. Pew Research Center. Internet/Broadband Fact Sheet. 2020; https://www.pewresearch.org/internet/fact-sheet/mobile/. Accessed January 25, 2021.

#### 5 PROTOCOL SIGNATURE PAGE

**Protocol Title**: Community-Centered Interventions for Improving Vaccine Uptake for COVID-19: Getting to Yes, Michigan!

Protocol Number: Version 12.0

Protocol Version/ Date: February 26, 2024

Sponsor Name: National Institutes of Health

# **Declaration of Investigator**

I confirm that I have read the above-mentioned protocol and its attachments. I agree to conduct the described trial in compliance with all stipulations of the protocol, regulations and ICH E6 Guideline for Good Clinical Practice (GCP).

Principal Investigator Name: Ken Resnicow, Ph.D.

Principal Investigator Signature:

Date: 2/26/24